CLINICAL TRIAL: NCT05804071
Title: Analysis of the Effect of Different Doses, Frequencies and Ways of Iron Supplements on Iron Deficiency Anemia in Pregnancy: a Randomized , Single Centered，Controlled, Single-blind Trial
Brief Title: Analysis of the Effect of Iron Supplements on Iron Deficiency Anemia in Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXL-KY-2023（006）
Record Dates: First submitted 2023-03-02; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Iron Deficiency Anemia of Pregnancy; Iron Storage Disease
MeSH Terms: conditions — Hemochromatosis | interventions — Niferex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 150mg QD (Active Comparator): Each subject took vitamin C 1 tablet and 150mg polysaccharide iron complex at 20:00 ± 1 hour every day.
  Interventions: Drug: Niferex
- 150mg QOD (Active Comparator): Each subject took vitamin C 1 tablet and 150mg polysaccharide iron complex at 20:00 ± 1 hour every other day.
  Interventions: Drug: Niferex
- 300mg QD (Active Comparator): Each subject took vitamin C 1 tablet and 300mg polysaccharide iron complex at 20:00 ± 1 hour every day.
  Interventions: Drug: Niferex
- 300mg QOD (Active Comparator): Each subject took vitamin C 1 tablet and 300mg polysaccharide iron complex at 20:00 ± 1 hour every other day.
  Interventions: Drug: Niferex
- Intravenous iron supplement (Active Comparator): Each subject was given intravenous iron supplements according to the instructions
  Interventions: Drug: Niferex

INTERVENTIONS:
Drug: Niferex — Daily iron supplement scheme (QD)：Oral polysaccharide iron complex capsule (Niferex)150mg/300mg daily.
  Alternative iron supplement scheme（QOD）：Oral polysaccharide iron complex capsule(Niferex) 150mg/300mg every other day.
  Intravenous iron supplement(MonoFer):use as instructions
  Other Names: MonoFer

SUMMARY:
Subjects were tested for hemoglobin, ferritin, serum iron, transferrin saturation and reticulocyte count during routine prenatal examination at 24-26 weeks of gestation, and blood samples were taken for serum hepcidin detection in the laboratory and the values were recorded. Those who met the criteria were included in the study group, signed the informed consent form and randomized into groups, and were given different drug administration schemes (150mg orally every day, 300mg orally every day, 150mg orally every other day, 300mg orally every other day, intravenous). At the same time, each subject was given anemia diet education, and all subjects were given folic acid 400ug/d and vitamin C 0.5g/d orally during the treatment period. If the subjects were in the oral iron group, the same time of oral iron was determined as 20 o'clock ± 1 hour in the evening, and the oral iron was not taken with other drugs; If the subject is in the intravenous medication group, the medication is scheduled to be administered at a uniform time of 8 o'clock ± 1 hour in the morning. The above subjects were followed up. Hemoglobin, ferritin, serum iron, transferrin saturation and reticulocyte count were performed at 30-32 and 37 weeks of pregnancy and delivery, and blood samples were taken for serum hepcidin detection in the laboratory and the values were recorded. The adverse reactions were investigated with a questionnaire at the last prenatal examination before delivery. After full term delivery, the patient fills in the delivery information and enters it into the database. Finally, the data statistician and the above personnel used the blind method for statistical analysis and reached a conclusion.

DETAILED DESCRIPTION:
Subjects were tested for hemoglobin, ferritin, serum iron, transferrin saturation and reticulocyte count during routine prenatal examination at 24-26 weeks of gestation, and blood samples were taken for serum hepcidin detection in the laboratory and the values were recorded. Those who met the criteria were included in the study group, signed the informed consent form and randomized into groups, and were given different drug administration schemes (150mg orally every day, 300mg orally every day, 150mg orally every other day, 300mg orally every other day, intravenous). At the same time, each subject was given anemia diet education, and all subjects were given folic acid 400ug/d and vitamin C 0.5g/d orally during the treatment period. If the subjects were in the oral iron group, the same time of oral iron was determined as 20 o'clock ± 1 hour in the evening, and the oral iron was not taken with other drugs; If the subject is in the intravenous medication group, the medication is scheduled to be administered at a uniform time of 8 o'clock ± 1 hour in the morning. The above subjects were followed up. Hemoglobin, ferritin, serum iron, transferrin saturation and reticulocyte count were performed at 30-32 and 37 weeks of pregnancy and delivery, and blood samples were taken for serum hepcidin detection in the laboratory and the values were recorded. The adverse reactions were investigated with a questionnaire at the last prenatal examination before delivery. After full term delivery, the patient fills in the delivery information and enters it into the database. Finally, the data statistician and the above personnel used the blind method for statistical analysis and reached a conclusion.

1.1 Oral iron：NIFEREX®（Each granule contains 0.15g of polysaccharide iron complex ，Kremers Urban Pharmaceuticals Inc.

） 1.2 Daily iron supplement scheme (QD)：Oral polysaccharide iron complex capsule 150mg/300mg daily.

1.3 Alternative iron supplement scheme（QOD）：）Oral polysaccharide iron complex capsule 150mg/300mg every other day 2.1Intravenous iron supplement：Iron Isomaltoside Injection（5ml： 500mg，Wasserburger Arzneimittelwerk GmbH）,Intravenous iron supplement

ELIGIBILITY:
Inclusion Criteria:

* The patient was examined and delivered at the First Affiliated Hospital of Shandong First Medical University (Qianfo Mountain Hospital of Shandong Province)
* Clinical diagnosis of ID（iron depletion）
* Clinical diagnosis of IDA（iron depletion anemia）
* In the second trimester of pregnancy (24-26 weeks of pregnancy)
* Must be able to swallow tablets
* Agree to participate in the trial and sign the informed consent.

Exclusion Criteria:

* C-reactive protein in serum ≥5mg/L；
* Clinical diagnosis of Hypertensive disorders complicating pregnancy
* Clinical diagnosis of Gestational diabetes
* Clinical diagnosis of Hypothyroidism
* Clinical diagnosis of Chronic digestive system diseases
* Clinical diagnosis of Renal insufficiency
* Clinical diagnosis of psychiatric diseases
* Clinical diagnosis of fetal growth restriction
* Clinical diagnosis of placenta previa
* Clinical diagnosis of placental abruption
* Clinical diagnosis of fetal distress
* Clinical diagnosis of premature rupture of membranes
* Clinical diagnosis of Thalassemia
* Clinical diagnosis of Hemoglobinopathy
* Use anticoagulant drugs for treatment
* Smoking
* Excessive drinking
* Clinical diagnosis of Hemorrhoids
* Take acid inhibitor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of childbearing age who can be pregnant
Enrollment: 452 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Ferritin | 37-41 weeks gestation
  Concentration of Ferritin in serum in late pregnancy
Elevated hemoglobin value | 37-41 weeks gestation
  Elevated hemoglobin value between 24 and 41 weeks of gestation

SECONDARY OUTCOMES:
Hemoglobin | 20-24 weeks gestation，30-32 weeks gestation，37-41 weeks gestation
  Concentration of Hemoglobin value in whole blood
ferritin | 20-24 weeks gestation，30-32 weeks gestation，37-41 weeks gestation
  Concentration of ferritin value in serum
serum iron | 20-24 weeks gestation，30-32 weeks gestation，37-41 weeks gestation
  Concentration of serum iron value in serum
transferrin saturation | 20-24 weeks gestation，30-32 weeks gestation，37-41 weeks gestation
  Concentration of transferrin saturation value in serum
total iron binding force | 20-24 weeks gestation，30-32 weeks gestation，37-41 weeks gestation
  total iron binding force in serum
reticulocyte count | 20-24 weeks gestation，30-32 weeks gestation，37-41 weeks gestation
  reticulocyte count in whole blood
Correction rate of iron deficiency anemia during pregnancy | 37-41 weeks gestation
  Correction rate of ferritin deficiency
Adverse reaction rate | 37-41 weeks gestation
  Rate of Adverse reaction such as Vomiting, nausea, constipation, diarrhea or allergy
Correction rate of ferritin deficiency | 37-41 weeks gestation
  Correction rate of ferritin deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Zhiwei, PH.D, Study Chair — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China